CLINICAL TRIAL: NCT02052401
Title: Domiciliary Intervention by Occupational Therapy After Hospital Discharge, to Prevent Rehospitalization in Elderly: Randomized Clinical Trial
Brief Title: Domiciliary Intervention by Occupational Therapy to Prevent Elderly Rehospitalization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Gerardo F Fasce Pineda, MD, Medical Doctor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SA13I20184
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Rehospitalization
Keywords: OLD AGE; Elderly; Domiciliary Intervention; Occupational Therapy; Rehospitalization

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Occupational Therapy Intervention (Experimental): Post Discharge Domiciliary Intervention by Occupational Therapy (OT)
  Interventions: Other: Domiciliary Intervention
- Usual follow-up (No Intervention): Usual follow-up of post discharge elderly patients, including pharmacological, and non-pharmacological care.

INTERVENTIONS:
Other: Domiciliary Intervention — Two time domiciliary application of an standardized protocol consisting of: a) evaluation of pharmacological and non pharmacological therapies adherence. b) application of a Checklist of home safety measures. c) development of a patient oriented occupational routine d) education in strategies for elderly global stimulation e) education strategies for identifying red flags and for correct use of health services.
  Arms: Occupational Therapy Intervention

SUMMARY:
The purpose of this study is to determine whether a home visit by an Occupational Therapist is effective in reducing the rehospitalization rates in elderly patients after hospital discharge.

DETAILED DESCRIPTION:
Introduction: The hospitalization of the elderly is a frequent event that is associated with complications including loss of functionality, which makes it difficult for the person to reinstate to their original context after discharge, increasing the likelihood of rehospitalization.

Objective : To describe and compare the impact of home-based intervention by Occupational Therapists (OT) in the likelihood of rehospitalization at 6 months versus usual care in persons older than 60 years after discharge.

Design : Randomized controlled trial in medical units of the Hospital Clínico de la Universidad de Chile (HCUCh) and Hospital de la Fuerza Aérea de Chile (HFACH)

Patients: Two hundred and six patients aged 60 years or older admitted for acute or decompensated chronic disease to either HCUCH or HFACH, with a life expectancy greater than 6 months, not institutionalized prior to hospitalization or discharge destination , and provided that they have a person of reference after hospital discharge .

Methods: The control group consists of the usual care regarding post discharge patients, in comparison to the experimental group, which , besides the usual discharge plan, considers a home visit from OT on 2 occasions for 6 months, who will apply the following plan of action: Compliance assessment of pharmacological and non-pharmacological indications, applying a checklist of home safety evaluation and structuring of an occupational routine, education of stimulation strategies, education in recognition of warning signs and proper use of health services. Patients will be recruited between 24 and 48 hours prior to hospital discharge where they will be invited to participate. Informed consent will be retrieved, and demographic information of patients and pre- hospitalization functional backgrounds will be collected during this period, and at discharge by means of Barthel Index (independence / dependence in basic activities of daily living (ADL)), Lawton & Brody Scale (ADL instrumental), Questionnaire Pfeffer Functional Activities ( FAQ), Confusion Assessment Method (CAM) (delirium at discharge), Pfeiffer Questionnaire (Short Portable Mental Status Questionnaire: SPMSQ ) (cognition), and Geriatrics Cumulative Illness Rating Scale disease ( CIRS -G) (comorbidity). Both groups will receive telephone follow-up at 4, 12 and 24 weeks after hospital discharge with intent to evaluate functionality and rehospitalization. Allocators, medical team giving hospital discharge, pone interviewers, and data analysts will be blind of the intervention allocation.

Expected Results: the home-based intervention after discharge with OT reduce the rate of rehospitalization in at least 40 % at 6 months in people over 60 years compared with usual care .

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* Living close by to domiciliary intervention occupational therapy team
* Hospitalised in Medical Unit for acute illness or complicated chronic disease
* Presence of a reference individual, over 18 years old, able to understand recommendations, with contact telephone number, and that shares SPENDS at least 20 hours with patient.
* Signed informed consent by patient

Exclusion Criteria:

* Estimated survival under 6 months
* Previous Institutionalisation or defined at discharge
* Reference individual with severe hearing problems that could interfere with telephone communication

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Rehospitalization Rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Fasce, MD, Principal Investigator — University of Chile
Locations (2):
- Chile (2):
  - Hospital Clinico de la Universidad de Chile, Santiago, Santiago Metropolitan
  - Hospital Fuerza Aérea de Chile, Santiago